CLINICAL TRIAL: NCT01731925
Title: A RANDOMIZED PHASE II DOUBLE-BLIND TRIAL OF SUNITINIB VERSUS PLACEBO IN COMBINATION WITH LANREOTIDE IN PATIENTS WITH PROGRESSIVE ADVANCED/METASTATIC MIDGUT CARCINOID TUMORS
Brief Title: A Study of Sunitinib Versus Placebo in Combination With Lanreotide in Patients With Progressive Advanced/Metastatic Midgut Carcinoid Tumors
Acronym: SUNLAND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Pfizer (Industry); Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUNLAND D12-01; 2012-001098-94 (EudraCT Number)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Carcinoid Tumors
Keywords: midgut carcinoid tumors; progressive; advanced; metastatic
MeSH Terms: conditions — Carcinoid Tumor; Neoplasm Metastasis | interventions — lanreotide; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunitinib (Experimental): Sunitinib 37.5 mg daily. Lanreotide at the dose of 120 mg will be injected every 28 days as the reference treatment to control the carcinoid syndrome in both arms.
  Interventions: Drug: Lanreotide; Drug: Sunitinib
- Placebo (Placebo Comparator): Placebo (for sunitinib). Lanreotide at the dose of 120 mg will be injected every 28 days as the reference treatment to control the carcinoid syndrome in both arms.
  Interventions: Drug: Lanreotide; Drug: Placebo (for sunitinib)

INTERVENTIONS:
Drug: Lanreotide — Lanreotide at the dose of 120 mg will be injected every 28 days as the reference treatment to control the carcinoid syndrome in both arms.
Drug: Placebo (for sunitinib)
  Arms: Placebo
Drug: Sunitinib — Sunitinib 37.5 mg daily
  Arms: Sunitinib

SUMMARY:
Sunitinib may provide an opportunity for a novel therapeutic strategy for the treatment of subjects with neuroendocrine tumors.

DETAILED DESCRIPTION:
With the exception of surgery for localized disease, there is presently a lack of available therapies with proven survival benefit for patients with neuroendocrine tumors (NET). Available treatment options for unresectable disease include the use of somatostatin analogs, which may relieve symptoms related to hormonal hypersecretion. The efficacy of cytotoxic chemotherapy in patients with metastatic carcinoid tumors is also limited. Combinations of either streptozocin and cyclophosphamide, or streptozocin and 5-fluorouracil, appear to be inactive, and both regimens are associated with substantial toxicity.

Receptor tyrosine kinases (RTKs) are implicated in deregulated/ autocrine proliferation and survival of solid and hematologic cancer cells. Sunitinib malate is an orally administered small molecule that inhibits the tyrosine kinase enzymatic activities of the receptors for VEGF and PDGF, and also blocks signalling through the KIT, FLT3 and RET pathways.

Therefore, sunitinib malate may provide an opportunity for a novel therapeutic strategy for the treatment of subjects with NET.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with midgut well-differentiated Grade 1-2 endocrine tumor.
2. Local, locally advanced or metastatic disease documented as progressive by RECIST v1.1. on CT-scan or MRI at baseline and within 12 months prior to baseline.
3. 5HIAA levels superior to 1.5ULN as measured in each individual centre.
4. Disease that is not amenable to surgery with curative intent.
5. Presence of at least one measurable target lesion for further evaluation according to RECIST v1.1
6. Adequate organ function
7. ECOG Performance status 0 or 1.
8. Life expectancy superior or equal to 3 months.
9. Age superior or equal to 18 years.
10. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment. Breast feeding is not allowed. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
11. Able to swallow oral compound.
12. Signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial prior to enrollment.
13. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
14. Registration in a national health care system (CMU included).

Exclusion Criteria:

1. Patients with undifferentiated, poorly differentiated gastrointestinal neuroendocrine tumors, pancreatic neuroendocrine tumors, bronchial carcinoid tumors.
2. Patients with carcinoid tumors with the presence of an obstructive intestinal tumor.
3. Patients with uncontrolled cardiac complication as part of their carcinoid syndrome.
4. Current treatment with any chemotherapy, chemoembolization therapy, immunotherapy, or investigational anticancer agent
5. Current treatment with dose superior or equal to 120 mg per month of lanreotide
6. Prior treatment with any tyrosine kinase inhibitors or anti-VEGF angiogenic inhibitors. Prior treatment with non-VEGF-targeted angiogenic inhibitors such as everolimus or temsirolimus is permitted.
7. Patients who stopped everolimus treatment was less than 4 weeks prior to randomization.
8. Patients with concomitant treatment with interferon.
9. Patients previously treated with chemotherapy, loco-regional therapy (e.g., chemoembolization) or interferon with last administration less than 6 weeks prior to randomization or with toxicity not resolved to less or equal grade 1 at randomization.
10. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri.
11. Treatment with potent CYP3A4 inhibitors and inducers within 7 and 12 days, respectively prior to study drug administration.
12. Concomitant treatment with therapeutic doses of anticoagulants
13. Concomitant treatment with a drug having proarrhythmic potential
14. Unstable systemic diseases including uncontrolled hypertension or active uncontrolled infections.
15. Current treatment on another clinical trial.
16. Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
17. Ongoing cardiac dysrhythmias of NCI CTC grade superior or equal to 2, atrial fibrillation of any grade, or prolongation of the QTc interval to more than 450 msec for males or more than 470 msec for females.
18. Symptomatic brain metastases, spinal cord compression, or new evidence of brain or leptomeningeal disease.
19. Left ventricular ejection fraction inferior or equal 50% as measured by either multigated acquisition scan or echocardiogram.
20. Positive test for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
21. Patients with complicated, untreated lithiasis of the bile ducts
22. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | time from date of randomization to first progression of disease (PD) or death for any reason in the absence of documented PD, assessed up to 3 years after the beginning of the study
  To evaluate the efficacy of the combination of sunitinib malate with lanreotide acetate and of placebo with lanreotide acetate regarding progression-free-survival (PFS) as assessed by the investigator, in patients suffering from progressive, advanced/metastatic midgut carcinoid tumors.

SECONDARY OUTCOMES:
Overall survival (OS) | time from date of randomization to date of death, assessed up to 3 years after the beginning of the study
  To evaluate overall survival (OS) in sunitinib- and placebo-treated subjects.
Objective response (OR) | from randomization until disease progression, assessed up to 3 years after the beginning of the study
  To evaluate objective response (OR) rate in sunitinib- and placebo-treated subjects.
Duration of response (DR) | time from CR or PR to objective tumor progression or to death due to any cause, whichever occurs first, assessed up to 3 years after the beginning of the study
  To evaluate duration of response (DR) in sunitinib- and placebo-treated subjects in subjects achieving a response.
Time to tumor response (TTR) | time from date of randomization to first documentation of objective tumor response that is subsequently confirmed.assessed up to 3 years after the beginning of the study
  To assess time to tumor response (TTR) for sunitinib- and placebo-treated subjects.
Biological responses | from baseline to end of treatment, assessed up to 3 years after the beginning of the study
  To evaluate the best biological responses as assessed using serum chromogranin A and urine 5HIAA for sunitinib- and placebo-treated subjects.
Safety | from visit 1 to 1 month after last study drug administration, assessed up to 3 years after the beginning of the study
  To assess safety and tolerability of sunitinib in the study population.
Quality of life | From screening to 1 month after last study drug administration, assessed up to 3 years after the beginning of the study
  To assess Health related Quality of life (EORTC QLQ C-30).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal HAMMEL, MD, Principal Investigator — Hôpital Beaujon
Locations (20):
- Belgium (6):
  - Cliniques Universitaires Saint Luc, Brussels
  - Institut Jules Bordet, Brussels
  - ULB Erasme, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- France (14):
  - Hôpital Saint André, Bordeaux
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Hopital Saint Vincent de Paul, Lille
  - Hôpital Edouard Herriot, Lyon
  - CHU La Timone, Marseille
  - Hôpital St Antoine, Paris
  - CHU Cochin, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - CHU Rouen, Rouen
  - CHRU Trousseau, Tours